CLINICAL TRIAL: NCT02096380
Title: Randomized Trial of Comparing One Cycle With Three Cycles Induction Chemotherapy Using Docetaxel, Cisplatin and Fluorouracil in Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: The Value of Single-cycle TPF Induction Chemotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Tao Xu, Principal investigator, Department of radiation oncology for head and neck cancer, First People's Hospital of Foshan, First People's Hospital of Foshan
Other Study IDs: FSHNG-1110
Record Dates: First submitted 2011-11-13; First posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; cycle; induction chemotherapy; docetaxel
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — neodymium pyrocatechin disulfonate; Induction Chemotherapy; Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- one cycle induction chemotherapy: Drug: docetaxel, cisplatin and fluorouracil
  Patients receive docetaxel (60mg/m2 on day 1), cisplatin (20mg/m2 on day 1-4) and fluorouracil (800mg/m2/d, continuous infusion, d1-4) every three weeks for single one cycle before the radiotherapy, then receive radical radiotherapy with IMRT and cisplatin (30mg/m2) every week for six cycles during radiotherapy.
  Other Names:
  docetaxel, cisplatin and fluorouracil
  Interventions: Drug: One cycle TPF induction chemotherapy for NPC
- three cycles induction chemotherapy: Drug: docetaxel, cisplatin and fluorouracil
  Patients receive docetaxel (60mg/m2 on day 1), cisplatin (20mg/m2 on day 1-4) and fluorouracil (800mg/m2/d, continuous infusion, d1-4) every three weeks for three cycles before the radiotherapy, then receive radical radiotherapy with IMRT and cisplatin (30mg/m2) every week for six cycles during radiotherapy.
  Other Names:
  docetaxel, cisplatin and fluorouracil
  Interventions: Drug: Three cycles TPF induction chemotherapy for NPC

INTERVENTIONS:
Drug: One cycle TPF induction chemotherapy for NPC — One cycle TPF induction chemotherapy for NPC
  Patients receive docetaxel (60mg/m2 on day 1), cisplatin (20mg/m2 on day 1-4) and fluorouracil (800mg/m2/d, continuous infusion, d1-4) every three weeks for single one cycle before the radiotherapy, then receive radical radiotherapy with IMRT and cisplatin (30mg/m2) every week for six cycles during radiotherapy.
  A total dose of 70Gy in 30 fraction to PTV-P, 60Gy in 30 fraction to PTV-1 and 54Gy in 30 fraction to PTV-2.
  Other Names: One cycle; induction chemotherapy; Docetaxel,; cisplatin; and 5-Fu
  Groups: one cycle induction chemotherapy
Drug: Three cycles TPF induction chemotherapy for NPC — Three cycles TPF induction chemotherapy for NPC
  Patients receive docetaxel (60mg/m2 on day 1), cisplatin (20mg/m2 on day 1-4) and fluorouracil (800mg/m2/d, continuous infusion, d1-4) every three weeks for three cycles before the radiotherapy, then receive radical radiotherapy with IMRT and cisplatin (30mg/m2) every week for six cycles during radiotherapy.
  A total dose of 70Gy in 30 fraction to PTV-P, 60Gy in 30 fraction to PTV-1 and 54Gy in 30 fraction to PTV-2.
  Other Names: Three cycles; induction chemotherapy; Decotaxel,; Cisplatin; and 5-Fu
  Groups: three cycles induction chemotherapy

SUMMARY:
Two Phase Ⅲ trials (TAX323 and TAX324) showed induction chemotherapy adding docetaxel to cisplatin plus fluorouracil (TPF) could significant improve survival in head and neck cancer, and a Phase Ⅱ trial from Hong Kong by Hui and colleges with this strategy has also been reported in nasopharyngeal carcinoma (NPC). However, whether three cycles induction could delay the whole time of treatment and reduce the survival benefit are still unknown. A retrospective study of one cycle TPF induction chemotherapy by the investigators group (not yet published) could improve survival in NPC. It encourage us to conduct this clinical trial.

DETAILED DESCRIPTION:
Patients presented with non-keratinizing NPC and stage Ⅲ-Ⅳb T3-4N1M0/TxN2M0 are randomly assigned to receive one cycle induction chemotherapy (docetaxel+cisplatin+fluorouracil) plus concurrent chemoradiotherapy (investigational arm) or three cycles induction chemotherapy (docetaxel+cisplatin+fluorouracil) plus concurrent chemoradiotherapy (investigational arm)(control arm). Patients in both arms receive radical Intensity modulated radiation therapy (Trilogy, Varian), and cisplatin (30mg/m2) every weeks for six cycles during radiotherapy. Radiation is delivered to GTV at 70 Gy in 30 fractions, CTV1 at at 60 Gy in 30 fractions and CTV2 at 54 Gy in 30 fractions. Patients in the investigational arm receive docetaxel (60mg/m2 on day 1), cisplatin (20mg/m2 on day 1-4) and fluorouracil (800mg/m2/d,continuous infusion, day 1-4) every three weeks for one cycle or three cycles before the radiotherapy. The primary end point is response rates after radiotherapy, failure-free survival (FFS) and toxic effects and treatment compliance. Secondary end points include overall survival (OS), distant failure-free survival (D-FFS), locoregional failure-free survival (LR-FFS). All efficacy analyses are conducted in the intention-to-treat population; the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing (according to World Health Organization (WHO 2005) histologically type).
* Satisfactory performance status: Karnofsky scale (KPS) > 70.
* Tumor staged is according to the 7th American Joint Commission on Cancer edition as Stage III：T1-2N2M0, T3N0-2M0 Stage IVa：T4N0-2M0
* Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.
* Adequate renal function: creatinine clearance ≥60 ml/min.

Exclusion Criteria:

* Age >60 years or <18 years.
* Pregnancy or lactation.
* Treatment with palliative intent.
* Prior radiotherapy, chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease including unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control and emotional disturbance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with locoregionally advanced nasopharyngeal carcinoma and agree to receive anti-cancer treatment in our hospital
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 3 year
  Failure-free survival is calculated from the date of randomization to the date of the first failure at any site.

SECONDARY OUTCOMES:
Locoregional failure-free survival | 3-year
  the data of randomization to the first local failure,
Overall survival | 3-year
  Overall survival is calculated from randomization to death from any cause.
Distant failure-free survival | 3-year
  the data of randomization to the first remote failure

CONTACTS AND LOCATIONS:
Overall Officials: Hong W Wei, M.D., Study Director — First People's Hospital of Foshan

REFERENCES:
- [Background] Kurita H, Yamamoto E, Nozaki S, Wada S, Furuta I, Miyata M, Kurashina K. Multicenter phase 2 study of induction chemotherapy with docetaxel and nedaplatin for oral squamous cell carcinoma. Cancer Chemother Pharmacol. 2010 Feb;65(3):503-8. doi: 10.1007/s00280-009-1056-z. Epub 2009 Jul 5. PMID 19579024
- [Background] Yoshioka T, Sakayori M, Kato S, Chiba N, Miyazaki S, Nemoto K, Shibata H, Shimodaira H, Ohtsuka K, Kakudo Y, Sakata Y, Ishioka C. Dose escalation study of docetaxel and nedaplatin in patients with relapsed or refractory squamous cell carcinoma of the esophagus pretreated using cisplatin, 5-fluorouracil, and radiation. Int J Clin Oncol. 2006 Dec;11(6):454-60. doi: 10.1007/s10147-006-0610-5. Epub 2006 Dec 25. PMID 17180514
- [Background] Janinis J, Papadakou M, Panagos G, Panousaki A, Georgoulias V, Hatzidaki D, Lefantzis D, Dokianakis G. Sequential chemoradiotherapy with docetaxel, cisplatin, and 5-fluorouracil in patients with locally advanced head and neck cancer. Am J Clin Oncol. 2001 Jun;24(3):227-31. doi: 10.1097/00000421-200106000-00003. PMID 11404490
- [Background] Hui EP, Ma BB, Leung SF, King AD, Mo F, Kam MK, Yu BK, Chiu SK, Kwan WH, Ho R, Chan I, Ahuja AT, Zee BC, Chan AT. Randomized phase II trial of concurrent cisplatin-radiotherapy with or without neoadjuvant docetaxel and cisplatin in advanced nasopharyngeal carcinoma. J Clin Oncol. 2009 Jan 10;27(2):242-9. doi: 10.1200/JCO.2008.18.1545. Epub 2008 Dec 8. PMID 19064973
- [Background] Lorch JH, Goloubeva O, Haddad RI, Cullen K, Sarlis N, Tishler R, Tan M, Fasciano J, Sammartino DE, Posner MR; TAX 324 Study Group. Induction chemotherapy with cisplatin and fluorouracil alone or in combination with docetaxel in locally advanced squamous-cell cancer of the head and neck: long-term results of the TAX 324 randomised phase 3 trial. Lancet Oncol. 2011 Feb;12(2):153-9. doi: 10.1016/S1470-2045(10)70279-5. Epub 2011 Jan 11. PMID 21233014
- [Background] Posner MR, Hershock DM, Blajman CR, Mickiewicz E, Winquist E, Gorbounova V, Tjulandin S, Shin DM, Cullen K, Ervin TJ, Murphy BA, Raez LE, Cohen RB, Spaulding M, Tishler RB, Roth B, Viroglio Rdel C, Venkatesan V, Romanov I, Agarwala S, Harter KW, Dugan M, Cmelak A, Markoe AM, Read PW, Steinbrenner L, Colevas AD, Norris CM Jr, Haddad RI; TAX 324 Study Group. Cisplatin and fluorouracil alone or with docetaxel in head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1705-15. doi: 10.1056/NEJMoa070956. PMID 17960013
- [Background] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012